CLINICAL TRIAL: NCT01470404
Title: Pharmacogenomic Study to Predict Toxicity and Response in Gastric Cancer Patients Treated With Adjuvant Chemotherapy
Brief Title: Pharmacogenomic Study (Adjuvant Chemotherapy)
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Ki Kang, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Other Study IDs: 2008-05-053
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adjuvant chemotherapy: Patients enrolled on to the adjuvant XP trial + patients who received adjuvant chemotherapy following curative resection of gastric cancer

SUMMARY:
To assess the role of germline polymorphisms in xenobiotic metabolism genes in toxicity profile.

To assess the role of germline polymorphisms in genes associated with DNA repair, p53 tumor suppressor gene and angiogenesis pathway in predicting recurrence and survival in gastric cancer patients treated with adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* gastric cancer patients treated with adjuvant chemotherapy

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on to the adjuvant trial will be considered as candidates for the study. Once the patient signed written informed consent, 10cc blood will be drawn in EDTA tube for DNA extraction.
Sampling Method: Probability Sample
Enrollment: 792 (Actual)
Dates: Start 2008-07-10 (Actual); Primary Completion 2013-05-10 (Actual); Study Completion 2013-07-10 (Actual)

PRIMARY OUTCOMES:
germline polymorphisms in xenobiotic metabolism genes in toxicity profile | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: won ki kang, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea